CLINICAL TRIAL: NCT01417104
Title: Aliskiren Effect on Plaque Progression In Established Atherosclerosis Using High Resolution 3D MRI (ALPINE): A Double Blind Placebo Controlled Trial
Brief Title: Aliskiren Effect on Aortic Plaque Progression
Acronym: ALPINE
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Safety concerns with approved medication identified in an unrelated trial
Sponsor: Ohio State University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSPP100AUS33T; NCT01123629 (obsolete NCT alias)
Record Dates: First submitted 2011-08-08; First posted 2011-08-16 (Estimated); Results first posted 2012-12-31 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Atherosclerosis
Keywords: plaque; magnetic resonance imaging (MRI); high blood pressure; MI; heart attack; CVA; stroke; PAD
MeSH Terms: conditions — Atherosclerosis; Plaque, Amyloid; Hypertension; Myocardial Infarction; Stroke | interventions — aliskiren; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aliskiren (Active Comparator): Aliskiren will be administered for 2 weeks at 150mg/day oral pill, followed by 34 weeks oral therapy with 300mg/day
  Interventions: Drug: Aliskiren
- Placebo (Placebo Comparator): Placebo (sugar pill) built to mimic both the 150mg Aliskiren tablet ( administered for the first 2 weeks) and the 300mg Aliskiren tablet ( administered for the rest of treatment period)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aliskiren — 150 mg/300mg
  Other Names: Tekturna
  Arms: Aliskiren
Drug: Placebo — 150mg/300mg
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
This study is being done to assess the effectiveness of short term (~9 months) Aliskiren/Placebo therapy to slow down the progression of atherosclerotic disease in thoracic and abdominal aorta. This will be checked by comparing before and after therapy magnetic resonance imaging (MRI) pictures of the aortic wall. Aliskiren is an FDA approved drug for hypertension but in this study is used for a new indication. Recent studies with animals have shown that Aliskiren therapy reduces the atherosclerotic plaque. Therefore, in this study, the investigators would like to evaluate whether the investigational drug Aliskiren, which is not FDA approved for this indication has the same beneficial effects in people with atherosclerotic disease.

DETAILED DESCRIPTION:
Treatments and Clinic Visits:

The 36-week double-blind, randomized treatment phase of the trial is preceded by 2-week single-blind placebo period to assess eligibility into the active treatment period, compliance, and to confirm the baseline blood pressure values of the enrolled subjects. If at the end of the single-blind phase, inclusion criteria will not be met, the participants will not be allowed to continue on to the trial. If they are eligible they will undergo baseline MRI studies after being randomized to either placebo or Aliskiren 150 mg, with an escalation to 300 mg at 2 weeks into treatment. This dose will be maintained for the duration of the trial. After randomization and dose escalation visits (at 2 weeks), patients will return for scheduled clinic visits at weeks 12 and 36. Assessment of routine safety measures including serum creatinine and potassium will be performed at pre-designated visits (randomization, drug escalation and end-of trial). At each study visit, after having the patient in a sitting position for 5 minutes, SBP/diastolic blood pressure will be measured 3 times in accordance with the AHA Committee Report on blood pressure determination. The patient will be then asked to stand for 2 minutes, and a single blood pressure measurement will be measured in the standing position. Evidence of left ventricular hypertrophy (LVH) will be determined using the Romhilt-Estes scoring system at baseline. Specialized measurements of plasma including insulin, glucose measures, adipokines (leptin and adiponectin) and high- sensitivity C-reactive protein (hsCRP) will be performed at randomization and 12 weeks into the trial. Central aortic blood pressure assessment will be performed at randomization and end of trial/exit visits (SphygmoCor CP, AtCor Medical, Itaska, Illinois, USA). Plasma direct renin measurements will be obtained at baseline and 12 weeks in part to assess compliance of patients with their therapy (Diasource, Belgium).

ELIGIBILITY:
Inclusion Criteria: Patients, both males and females, were eligible if they were ≥ 45 years of age, with previously documented cardiovascular disease, defined as at least one of the following: myocardial infarction (MI), cerebrovascular accident (CVA), coronary bypass surgery and/or percutaneous intervention, peripheral arterial disease (PAD), defined as ankle brachial index (ABI) <0.9 and/or prior peripheral intervention/surgery. Subjects on angiotensin-converting enzyme inhibitor (ACEI) or angiotensin receptor blockers (ARB) therapy were eligible to participate, provided no dose adjustments were made during the course of the study.

Exclusion Criteria: Contraindications to the MRI exam (pacemakers, metallic implants, severe claustrophobia); diagnosis of Type II Diabetes or use of hypoglycemic drugs; uncontrolled hypertension (>145/90 mm Hg); low density lipoprotein (LDL) of ≥ 130mg/dL; renal insufficiency defined as glomerular filtration rate (GFR) ≤ 40 ml/minute (derived by the Modified Diet in Renal Disease (MDRD) equation); initiation of new therapy with statins, ACEI/ARBs, anti-oxidants, calcium channel blockers, diuretics, β blockers; transient ischemic cerebral attack during the prior 6 months; history of allergy to renin inhibitors; unstable cardiac syndromes; symptomatic arrhythmias; history of malignancy including leukemia and lymphoma (but not basal cell skin cancer, cured squamous cell cancer and localized prostate cancer) and history of allergy to renin inhibitors.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Rajagopalan, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Derived] Deiuliis J, Mihai G, Zhang J, Taslim C, Varghese JJ, Maiseyeu A, Huang K, Rajagopalan S. Renin-sensitive microRNAs correlate with atherosclerosis plaque progression. J Hum Hypertens. 2014 Apr;28(4):251-8. doi: 10.1038/jhh.2013.97. Epub 2013 Oct 24. PMID 24152824
- [Derived] Mihai G, Varghese J, Kampfrath T, Gushchina L, Hafer L, Deiuliis J, Maiseyeu A, Simonetti OP, Lu B, Rajagopalan S. Aliskiren effect on plaque progression in established atherosclerosis using high resolution 3D MRI (ALPINE): a double-blind placebo-controlled trial. J Am Heart Assoc. 2013 May 17;2(3):e004879. doi: 10.1161/JAHA.112.004879. PMID 23686372

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from The Ohio State Medical Center and Columbus surrounding area between April 2009 to December 2011.
Pre-assignment Details: 187 participants screened; 116 did not meet inclusion criteria or meet exclusion criteria; 71 randomized.
Period: Overall Study
Arm/Group | Aliskiren | Placebo
Started | 34 | 37
Completed | 28 | 35
Not Completed | 6 | 2
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Failure to make contact | 0 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren | Placebo | Total
Number analyzed (Participants) | 34 | 37 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 13 | 30
  >=65 years | 17 | 24 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (11.5) | 64.5 (8.9) | 64.18 (10.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 12
  Male | 25 | 34 | 59
Region of Enrollment [Number; unit: participants]
  United States | 34 | 37 | 71

OUTCOME MEASURES:

1. Primary Outcome: Change in Normalized Total Aortic Wall Volume (TWV) Between the Trial Arms at the End of the Treatment
Description: All patients underwent imaging using a 3T, MRI system. The MRI sequence method used for wall depiction was a 3D, fat suppressed, dark blood, turbo spin echo sequence with variable flip angles (SPACE). Following co-registration of pre and post treatment MR images, and generation of MPR sections, images were magnified, contrast adjusted and patient/exam identifier information was removed and replaced by pre-assigned code to blind images for measurements.
  An experienced observer performed manual measurements of lumen and lumen plus wall areas by delineating the inner border and the outer border of the vessel wall in each cross-section image of the aorta. Using an approach similar to intravascular atheroma volume calculations, normalized total aortic wall volume (TWV) for thoracic region, abdominal region and total aorta for each patient and each exam was generated.
Time Frame: Baseline and end of treatment ( 17 to 36 weeks)
Population: 3 MRI data sets were not analyzable ( low quality images), and 23 post-treatment MRI not obtained ( <17 weeks on drug when trial terminated owing to ALTITUDE results)
Measure: Mean (Standard Deviation); unit: mm3
Groups:
- Aliskiren: Aliskiren was administered for 2 weeks at 150mg/day oral pill, followed by 34 weeks oral therapy with 300mg/day
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 18 | 19
mm3 | 5.31 (6.57) | 0.15 (4.39)
Statistical Analysis 1: Comparison: Aliskiren vs Placebo; Test type: Superiority or Other; p < 0.031, t-test, 2 sided; Mean Difference (Final Values) = 5.16, 95% CI 2-sided [0.85 to 9.47]

2. Secondary Outcome: Change in the Percentage Wall Volume (PWV) Between Baseline and End of Treatment
Description: Using an approach similar to intravascular atheroma volume calculations, percentage wall volume (PWV) for thoracic region, abdominal region and total aorta for each patient and each exam was generated. and a difference between baseline and end of treatment was calculated.
Time Frame: Baseline and end of treatment ( 17 to 36 weeks)
Population: 3 MRI not analyzable, 23 final MRI not obtained due to trial termination
Measure: Mean (Standard Deviation); unit: Percentage of the Outer Wall Volume
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 18 | 19
Percentage of the Outer Wall Volume | 3.37 (2.96) | 0.97 (2.02)
Statistical Analysis 1: Comparison: Aliskiren vs Placebo; Test type: Superiority or Other; p = 0.041, t-test, 2 sided; Mean Difference (Net) = 2.40, 95% CI 2-sided [0.44 to 4.36]

3. Other Pre Specified Outcome: Change From Baseline in Resting Diastolic Blood Pressure
Description: Difference between end of treatment and baseline in resting diastolic blood pressure
Time Frame: baseline to end of treatment ( up to 36 weeks)
Population: Intent to treat analysis including only participants who had at least one post-baseline assesment
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 28 | 35
mm Hg | -3.88 [-9.23 to 1.47] | -2.32 [-6.39 to 1.7]

ADVERSE EVENTS:
Time Frame: up to 36 weeks
Arm/Group | Aliskiren | Placebo
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/37
Other Adverse Events (participants affected / at risk) | 1/34 | 0/37
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aliskiren (N=34) | Placebo (N=37)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No